CLINICAL TRIAL: NCT06751407
Title: Comparison of Single-level and Two-level Serratus Posterior Superior Intercostal Plan Block (SPSIPB) Applications in the Treatment of Acute Pain After Mastectomy
Brief Title: Single-level and Two-level Serratus Posterior Superior Intercostal Plan Block (SPSIPB)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Seyyid Furkan Kına, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2024-0065
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-12

CONDITIONS: Opioid Consumption; Demographic Data
Keywords: serratus posterior superior intercostal plane block; pain; breast cancer; mastectomy
MeSH Terms: conditions — Pain; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Single level SPSIPB (Active Comparator): The procedure will be performed with the patient in the prone position in the preoperative period. After the scapula is slightly shifted laterally, the US probe is held sagittally at the upper corner of the scapula spine, and the 3rd rib and the serratus posterior superior muscle will be visualized. In plane technique will be used. The block needle will be advanced in the caudo-cranial direction and entered between the serratus posterior superior and the 3rd rib. The block location will be confirmed by injecting 2 ml of saline between the rib and the muscle. After the block location is confirmed, 20 ml of 0.25% bupivacaine will be used.
  Interventions: Procedure: Single level SPSIPB
- Group Two-level SPSIPB (Active Comparator): The block needle will be advanced in the caudo-cranial direction and inserted between the serratus posterior superior and the 2nd rib. The block location will be confirmed by injecting 2 ml of saline between the rib and the muscle. After the block location is confirmed, 10 ml of 0.25% bupivacaine will be used. Then, the US probe will be held sagittally in the medial part of the scapula spine, and the 4th rib and serratus posterior superior muscle will be visualized. In plane technique will be used. The block needle will be advanced in the caudo-cranial direction and inserted between the serratus posterior superior and the 4th rib. The block location will be confirmed by injecting 2 ml of saline between the rib and the muscle. After the block site is confirmed, 10 ml of 0.25% bupivacaine will be used. A total of 20 ml of 0.25% bupivacaine will be used.
  Interventions: Procedure: Two-level SPSIPB

INTERVENTIONS:
Procedure: Single level SPSIPB — The procedure will be performed with the patient in the prone position in the preoperative period. After the scapula is slightly shifted laterally, the US probe is held sagittally at the upper corner of the scapula spine, and the 3rd rib and the serratus posterior superior muscle will be visualized. In plane technique will be used. The block needle will be advanced in the caudo-cranial direction and entered between the serratus posterior superior and the 3rd rib. The block location will be confirmed by injecting 2 ml of saline between the rib and the muscle. After the block location is confirmed, 20 ml of 0.25% bupivacaine will be used.
  Arms: Group Single level SPSIPB
Procedure: Two-level SPSIPB — In plane technique will be used. The block needle will be advanced in the caudo-cranial direction and inserted between the serratus posterior superior and the 2nd rib. The block location will be confirmed by injecting 2 ml of saline between the rib and the muscle. After the block location is confirmed, 10 ml of 0.25% bupivacaine will be used. Then, the US probe will be held sagittally in the medial part of the scapula spine, and the 4th rib and serratus posterior superior muscle will be visualized. In plane technique will be used. The block needle will be advanced in the caudo-cranial direction and inserted between the serratus posterior superior and the 4th rib. The block location will be confirmed by injecting 2 ml of saline between the rib and the muscle. After the block site is confirmed, 10 ml of 0.25% bupivacaine will be used. A total of 20 ml of 0.25% bupivacaine will be used.
  Arms: Group Two-level SPSIPB

SUMMARY:
Breast cancer is the most common malignancy in women; one of the mainstays of breast cancer treatment is surgery, and modified radical mastectomy is one of the standard treatments. Postoperative pain can seriously reduce the quality of life in patients, and acute pain can even trigger chronic pain syndrome. Thoracic paravertebral, thoracic epidural, intercostal nerve, and interscalene brachial plexus blocks have been used for anesthesia and abrigation during modified radical mastectomy, but their applications are limited due to the complex nature of the procedures and serious complications. In recent years, regional nerve blocks, including intercostal nerve block, erector spinae plane block (ESPB), and paravertebral block, PECS I-II block, serratus anterior plane block (SAPB), and Serratus Posterior Superior Intercostal Plane Block (SPSIPB), have been applied for the treatment of postmastectomy pain in breast cancer patients. SPSIPB has been frequently used for the treatment of acute pain in the postoperative period following surgeries in the thoracic region. SPSIPB is placed on the spine of the scapula in the sagittal plane to identify the second and third ribs under USG guidance. After visualizing the trapezius and serratus posterior superior (SPS) by moving medially to the upper medial border of the scapula, a block is applied to the depths of the SPS from above the 3rd rib. The applied local anesthetic solution spreads under the SPS muscle. Ipsilateral postoperative analgesia is provided with SPSIPB. SPSIPB can be applied on the 3rd rib in one go, or on the 3rd and 4th ribs in two go. Thus, the local anesthetic solution can be distributed more effectively and more effective postoperative analgesia can be provided.

ELIGIBILITY:
Inclusion Criteria:

1-Those between the ages of 18-80

2.Those with ASA score I-II-III

3.Those with body mass index (BMI) between 18-40

4.Patients who underwent Single-Level or Two-Level SPSIPB together with mastectomy in the operating room

Exclusion Criteria:

1. Those under 18 and over 80
2. Those with ASA score IV and above
3. Those with advanced co-morbidities
4. Those with a history of bleeding diathesis
5. Patients with infection in the area where the block will be performed
6. Those with BMI under 18 and over 40
7. Patients who underwent surgery under emergency conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Intraoperative opioid consumption. | Intraoperative period
  Intraoperative opioid consumption will be recorded.

SECONDARY OUTCOMES:
Postoperative 24-hour numeric rating scale | postoperative 24 hours period
  Postoperative numeric rating scale will be recorded.(0: no pain-10: severe pain)

REFERENCES:
- [Background] Ciftci B, Alver S, Ahiskalioglu A, Bilal B, Tulgar S. Serratus posterior superior intercostal plane block for breast surgery: a report of three cases, novel block and new indication. Minerva Anestesiol. 2023 Nov;89(11):1054-1056. doi: 10.23736/S0375-9393.23.17432-3. Epub 2023 Jun 1. No abstract available. PMID 37272274
- [Background] Kulturoglu G, Altinsoy S, Ozguner Y, Cataroglu CK. Novel Serratus Posterior Superior Intercostal Plane Block Provided Satisfactory Analgesia after Breast Cancer Surgery: Two Case Reports. Turk J Anaesthesiol Reanim. 2024 Feb 28;52(1):33-35. doi: 10.4274/TJAR.2024.231431. PMID 38414179